CLINICAL TRIAL: NCT01707342
Title: A Phase I, Open-Label, Sequential, Single-Dose Study to Assess the Absolute Bioavailability and Pharmacokinetics of TMC435 Administered as Single Oral Doses of 50 mg and 150 mg and an Intravenous Microdose of 100 μg [3H]-TMC435 in Healthy Male Subjects
Brief Title: A Study to Assess the Absolute Bioavailability and Pharmacokinetics of Simeprevir (TMC435) Administered as Single Oral Doses of TMC435 and an Intravenous Microdose of [3H]-TMC435 in Healthy Male Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100901; TMC435-TiDP16-C118 (Other: Janssen R&D Ireland); 2012-002330-37 (EudraCT Number)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Male Participants
Keywords: Healthy male participants; Absolute bioavailability; Bioavailability; Pharmacokinetics; Simeprevir; TMC435; [3H]-TMC435; Hepatitis C virus; HCV
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Simeprevir (TMC435) (Experimental): Treatment A: single oral dose of simeprevir (TMC435) 50 mg; and Treatment B: single oral dose of simeprevir (TMC435) 150 mg. A single 10 minute intravenous infusion of [3H]-TMC435 (100 microcurie) 100 microgram will be followed 5 hours later after administration of Treatment A and Treatment B in Period 1 and Period 2, respectively.
  Interventions: Drug: Simeprevir (TMC435)

INTERVENTIONS:
Drug: Simeprevir (TMC435) — Treatment A: Simeprevir (TMC435) 50 mg; and Treatment B: Simeprevir (TMC435) 150 mg; will be followed 5 hours later by a single 10 minute intravenous infusion of [3H]-TMC435 (100 microcurie) 100 microgram in Period 1 and Period 2, respectively.

SUMMARY:
The purpose of this study is to evaluate the absolute bioavailability and pharmacokinetics (what the body does to the medication) of simeprevir (TMC435) after administration of single oral doses of 50 mg and 150 mg when administered together with a single intravenous (IV) dose of 100 microgram [3H]-TMC435 in healthy male participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), sequential (a single group of participants where study medication is administered in a sequence), single-dose study to assess the absolute bioavailability and pharmacokinetics (what the body does to the medication) of single oral doses of 50 mg and 150 mg simeprevir (TMC435) administered together with an intravenous (IV) microdose of 100 microgram [3H]-TMC435 in healthy male participants. The study consists of 3 phases, screening phase (21 days prior to administration of study medication), treatment phase, and a follow up phase. In the treatment phase, participants will receive 2 treatments, ie, Treatment A: single oral dose of simeprevir (TMC435) 50 mg followed 5 hours later by a single 10 minute IV infusion of [3H]-TMC435 (100 microcurie) 100 microgram; and Treatment B: single oral dose of simeprevir (TMC435) 150 mg followed 5 hours later by a single 10 minute IV infusion of [3H]-TMC435 (100 microcurie) 100 microgram. Treatments will be administered in two consecutive treatment periods, first Treatment A in Period 1, followed by Treatment B in Period 2; separated by a washout period (period when the participant is not receiving any study medication) of 7 to 14 days. The follow up will be for 5 to 7 days after end of Period 2. Blood samples will be collected for full plasma pharmacokinetics evaluations; along with urine and stool samples for analysis of total plasma radioactivity. Safety evaluations for adverse events, clinical laboratory tests, electrocardiogram, vital signs, physical examination, liver volume determination, and specific toxicities will be monitored throughout the study. The total duration of the study will be approximately 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram, and clinical laboratory tests performed at screening
* Must be non-smoking for at least 3 months prior to screening

Exclusion Criteria:

* History of liver or renal insufficiency
* Have any ferromagnetic medical implants or medical devices that can be de-programmed by strong magnetic fields such as, but not limited to: cardiac pacemakers, implantable cardiac defibrillators, cochlear implants, or insulin pumps
* Had a surgical intervention on brain or eyes or has an intraocular foreign metallic object
* Has a history of anxiety and claustrophobia

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of simeprevir (TMC435) | Pre-dose Day 1, post-dose Days 1-4
Volume of distribution of [3H]-TMC435 and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Maximum observed plasma concentration of simeprevir (TMC435), [3H]-TMC435, and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Time to reach the maximum observed plasma concentration of simeprevir (TMC435), [3H]-TMC435, and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Area under the concentration versus time curve from time of administration up to the last time point with a measurable concentration post dosing of simeprevir (TMC435), [3H]-TMC435, and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Area under the concentration versus time curve extrapolated to infinity of simeprevir (TMC435), [3H]-TMC435, and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Area under the first moment of the concentration versus time curve from the time of dosing up to a definite time, to infinity, or to the time of the last measureable concentration of [3H]-TMC435 and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Mean residence time of [3H]-TMC435 and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Terminal elimination rate constant of simeprevir (TMC435), [3H]-TMC435, and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Terminal elimination half-life of simeprevir (TMC435), [3H]-TMC435, and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4
Total systemic clearance of drug following single-dose intravenous administration of [3H]-TMC435 and [3H]-total radioactivity | Pre-dose Day 1, post-dose Days 1-4

SECONDARY OUTCOMES:
Total radioactivity excreted into the feces from time 0 to the time of discharge | Post-dose Hours 5, 24, 48, 72, and 96
Total radioactivity excreted into the feces expressed as a percentage of the administered dose | Post-dose Hours 5, 24, 48, 72, and 96
Total radioactivity excreted into urine from time 0 to the time of discharge | Post-dose Hours 5, 24, 48, 72, and 96
Total radioactivity excreted into the urine expressed as a percentage of the administered dose | Post-dose Hours 5, 24, 48, 72, and 96
Number of participants with adverse events | up to 30 days after dose of study medications

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Merksem, Belgium